CLINICAL TRIAL: NCT04184804
Title: A School-based Intervention Programme to Promote Organic Fruit and Vegetable Consumption in Primary School-children: A Cluster-randomized Feasibility Trial (PRISHEC)
Brief Title: Feasibility Trial on Organic Fruit and Vegetable Consumption in Primary School-children
Acronym: PRISHEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Konstantinos Makris, Dr. Konstantinos C. Makris, Associate Professor of Environmental Health, Cyprus University of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PRISHEC
Record Dates: First submitted 2019-11-27; First posted 2019-12-04 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Obesity
Keywords: organic; children; school; health promotion; fruits; vegetables
MeSH Terms: conditions — Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Intervention (Experimental): School-based intervention
  Interventions: Behavioral: Behavioral Intervention
- Control (No Intervention): Control. No intervention (usual education). The school does not receive any material and gets the information that they are part of a study on eating habits of primary school children.

INTERVENTIONS:
Behavioral: Behavioral Intervention — The intervention package will be consisted of:
  1. Introduction of organic fruits and vegetables (by replacing the conventional ones) in school lunch menus
  2. Signs in school areas about organic fruits and vegetables
  3. Workshops and interactive games for children
  4. Seminars for parents
  Arms: Behavioral Intervention

SUMMARY:
The aim of this trial is to examine the feasibility of a larger-scale intervention study (regional study in schools run by the Ministry of Education) to increase the consumption of fruits and vegetables in schools towards reducing percentages of childhood obesity prevalence rates by at least 0.5% every two years for all children, using an organic-based healthy eating intervention package for primary school children and their parents.

DETAILED DESCRIPTION:
Pre-implementation phase: All necessary approvals (Bioethics, Ministry of Education) for the implementation of the study will be taken. Initial contacts with school directors will be done to obtain their approval.

Preparatory phase: Contact with the parents' union will be done, to explain the aim of the study and bring them in contact with interested organic companies in order to reach an agreement for the cost of providing organic fruits and vegetables in school lunch menus. Following the agreement, parents and children will be informed about the study through separate seminars for children and parents and a flyer that will be sent at home. Signed consent forms will be obtained. Teachers will also be taken on board and information pertaining to the overall scope and objectives of the study will be shared with them. This phase will also involve pre-testing of all the data collection tools. After pre-testing, necessary modifications will be carried out in the tools.

Intervention phase: At the beginning of the intervention (March 2020), a baseline questionnaire with demographic data and a food frequency questionnaire (FFQ) to record the children's diet habits will be administered to parents. Organic fruits and vegetables will be introduced at the school lunch menu and one workshop for children will be implemented per month. The workshops will include interactive games for children. Signs will be posted in various school areas. At the end of the intervention (end of May 2020), a seminar for parents will take place in order to discuss their children's impression of the program. FFQ and evaluation questionnaires (feedback on the intervention) will be administered to parents.

For the control group: No intervention (usual education). School directors are contacted and their approval is requested to conduct the study that aims to assess the eating habits of primary school children. The parents will be informed about the study with a flyer that will be sent at home through school and signed informed consents will be obtained. A baseline questionnaire with demographic data and an ffq will be administered to parents about their children in March 2020. Another ffq will be administered at the end of May 2020.

ELIGIBILITY:
Inclusion Criteria:

* Primary school children attending the all-day school meals

Exclusion Criteria:

* No exclusion criteria are applied

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in reported consumption frequency of fruit and vegetables (organic and conventional) in children | baseline, 9 weeks
  Self-reported consumption of foods based on a food frequency questionnaire. This is based on the consumption frequency of food items for the last three months.

SECONDARY OUTCOMES:
Accrual rates | 9 weeks
  Number of participants recruited
Accrual losses | 9 weeks
  Number of participants declined/withdrawn to participate
Acceptability of the intervention by children (qualitative, proportions) | 9 weeks
  Use of an evaluation questionnaire on intervention acceptability, which will be administered to parents at the end of the intervention. This includes 4 closed and 4 open-ended questions.
Change in number of servings of fruits and vegetables consumed | 9 weeks
  Each teacher in charge during lunch period records the number of fruits and salad servings consumed (photos of non-consumed fruits and salad - 1 per week).
Change in reported consumption frequency of other food groups (meat and sweets/fats/oils groups) in children | baseline, 9 weeks
  Self-reported consumption of foods based on a food frequency questionnaire. This is based on the consumption frequency of food items for the last three months.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos C Makris, Principal Investigator — Cyprus University of Technology
Locations (1):
- Primary schools, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Upon publication, the IPD will be available through the journal's website
Supporting Information: Study Protocol
Time Frame: Upon publication of the study
Access Criteria: Publicly available

REFERENCES:
- [Background] Makris KC, Konstantinou C, Andrianou XD, Charisiadis P, Kyriacou A, Gribble MO, Christophi CA. A cluster-randomized crossover trial of organic diet impact on biomarkers of exposure to pesticides and biomarkers of oxidative stress/inflammation in primary school children. PLoS One. 2019 Sep 4;14(9):e0219420. doi: 10.1371/journal.pone.0219420. eCollection 2019. PMID 31483785
- [Background] Savva SC, Kourides YA, Hadjigeorgiou C, Tornaritis MJ. Overweight and obesity prevalence and trends in children and adolescents in Cyprus 2000-2010. Obes Res Clin Pract. 2014 Sep-Oct;8(5):e426-34. doi: 10.1016/j.orcp.2013.11.005. Epub 2013 Dec 8. PMID 25263832
- [Background] WHO-COSI, World Health Organisation - COSI report: http://www.euro.who.int/en/healthtopics/disease-prevention/nutrition/publications/2018/childhood-obesity-surveillance-initiative-cosifactsheet.-highlights-2015-17-2018